CLINICAL TRIAL: NCT04647604
Title: Resolving Inflammatory Storm in COVID-19 Patients by Omega-3 Polyunsaturated Fatty Acids - A Single-blind, Randomized, Placebo-controlled Feasibility Study
Brief Title: Resolving Inflammatory Storm in COVID-19 Patients by Omega-3 Polyunsaturated Fatty Acids -
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Magnus Bäck, Professor of Cardiology, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-002293-28
Record Dates: First submitted 2020-06-12; First posted 2020-12-01 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: Inflammatory Storm; COVID-19 infection; Omega-3 fatty acids; Inflammatory biomarkers; Omega-3 index
MeSH Terms: conditions — COVID-19 | interventions — fish oil triglycerides; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omega (Active Comparator): Omegaven® (2 mL/kg/day, equivalent to 6 g Docosahexaenoic Acid (DHA)+Eicosapentaenoic Acid (EPA) in a 70 kg individual) once daily for 5 days
  Interventions: Drug: Omegaven®
- Sodium chloride (NaCl) (Placebo Comparator): 2 mL/kg/day) once daily for 5 days
  Interventions: Drug: Sodium chloride

INTERVENTIONS:
Drug: Omegaven® — A highly refined fish oil in an emulsion for infusion with purified egg phosphatides and glycerol.
  Arms: Omega
Drug: Sodium chloride — intravenously administered 2 mL/kg/day
  Arms: Sodium chloride (NaCl)

SUMMARY:
A study on patients who are hospitalized and tested positive for COVID-19 or have a typical CT image of COVID-19 infection, to establish if omega-3 Polyunsaturated Fatty Acid (PUFA) supplementation by intravenous route is a possible treatment option in COVID-19 with minimal risks to the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed informed consent prior to any study specific procedures.
2. Female and male patients ≥18 years of age.
3. COVID-19 positive or typical CT image of COVID-19 infection.
4. Clinical status requiring hospitalization.

Exclusion Criteria:

1. According to Omegaven® contraindications (serious bleeding disorders, acute life-threatening condition, including acute shock, acute myocardial infarction, acute stroke, acute emboli, and coma).
2. Known hypersensitivity to Omegaven® or any of the ingredients.
3. Participation in any clinical research study evaluating an investigational medicinal product (IMP) within 3 months prior to screening.
4. Pregnancy and breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-07-07 (Actual)

PRIMARY OUTCOMES:
Changes in inflammatory biomarkers | 5 days
  white blood cell counts
Changes in inflammatory biomarkers | 5 days
  CRP
Changes in inflammatory biomarkers | 5 days
  lipidomic profiling
Changes in inflammatory biomarkers | 5 days
  cytokines
Changes in inflammatory biomarkers | 5 days
  metabolomic profiling

SECONDARY OUTCOMES:
Changes in proresolving mediators | 5 days
  lipidomics
Changes in fatty acids in the erythrocyte fraction | 5 days
  fatty acid profile
Changes in cardiac biomarkers | 5 days
  Troponin, NTproBNP
Changes in biomarkers of organ damage | 5 days
  LD, creatinine
Changes in thrombosis parameters | 5 days
  platelet count, D-dimer,
Changes in coagulation parameters | 5 days
  fibrinogen
Changes in markers of infection | 5 days
  procalcitonin concentrations
Changes in infection load | 5 days
  SARS-CoV2-RNAemia
Changes in clinical parameters | through study completion, on average 10 days
  National Early Warning Score (NEWS2)
Length of hospital stay | through study completion, on average 10 days
  Days of hospital stay
Complications | through study completion, on average 10 days
  ICU need, mortality

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Bäck, Professor, Principal Investigator — Karolinska University Hospital
Locations (2):
- Sweden (2):
  - Karolinska Universitetssjuhuset, Stockholm
  - Södersjukhuset, Stockholm

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported will be shared, after deidentification, with researchers who provide a methodologically sound proposal.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months following article publication and finishing 36 months following article publication.
Access Criteria: Study protocol will be published. Investigators interested in data should contact the principal investigator.

REFERENCES:
- [Derived] Arnardottir H, Pawelzik SC, Ohlund Wistbacka U, Artiach G, Hofmann R, Reinholdsson I, Braunschweig F, Tornvall P, Religa D, Back M. Stimulating the Resolution of Inflammation Through Omega-3 Polyunsaturated Fatty Acids in COVID-19: Rationale for the COVID-Omega-F Trial. Front Physiol. 2021 Jan 11;11:624657. doi: 10.3389/fphys.2020.624657. eCollection 2020. PMID 33505321